CLINICAL TRIAL: NCT00609427
Title: Effects of Cognitive Intervention for Older Adults With Memory Decline: A Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Lisa Koski, Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSY-07-015
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-06

CONDITIONS: Mild Cognitive Impairment
Keywords: cognitive training; cognitive rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- EA (Experimental): Training in external memory aids
  Interventions: Behavioral: External memory aids training
- MT (Experimental): Mnemonic training intervention
  Interventions: Behavioral: MEMO programme (Inst Universitaire de Geriatrie, Montreal)
- WL (No Intervention): Wait-list control

INTERVENTIONS:
Behavioral: MEMO programme (Inst Universitaire de Geriatrie, Montreal) — 8 weekly group training sessions in mnemonic strategies, administered by clinical psychologist.
  Arms: MT
Behavioral: External memory aids training — 8 weekly group sessions of training in the use of external memory aids, administered by clinical psychologist
  Arms: EA

SUMMARY:
The purpose of this study is to evaluate the effects of training in memory skills vs. use of external memory aids on everyday memory functioning in older people with mild cognitive impairment.

DETAILED DESCRIPTION:
Some older people experience memory loss that is worse than other people of their age, although they are not demented. This condition is known as mild cognitive impairment (MCI). Healthy older people can learn mnemonic strategies to improve their memory abilities. Can cognitive rehabilitation help people with MCI do better on mental tasks or maintain better functioning in everyday life? This study will evaluate the effects of two different rehabilitation programmes. Patients in the memory training group will learn mental strategies aimed at improving memory. Patients in the memory compensation group will learn to use external memory aids.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild cognitive impairment

Exclusion Criteria:

* Unable to speak and understand English
* Unable to comply with treatment program due to significant comorbid illness; OR
* Anticipated inability to attend all study sessions

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Rey Auditory Verbal Learning Test | 19-20 weeks
Wechsler Memory Scale - Logical Memory | 19-20 weeks
Face-name associations test | 19-20 weeks
Multifactorial Memory Questionnaire - Ability subscale | 19-20 weeks

SECONDARY OUTCOMES:
Rivermead Behavioural Memory Test | 19-20 weeks
FAS test (non-memory) | 19-20 weeks
Category fluency (non-memory test) | 19-20 weeks
Victoria Stroop Test (non-memory test) | 19-20 weeks
Digit Span (non-memory test) | 19-20 weeks
Multifactorial Memory Questionnaire - Strategies and Contentment subscales | 19-20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Koski, PhD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada